CLINICAL TRIAL: NCT04888650
Title: Assessment of the State of Health, Quality of Life and Expectations of Patients With Hereditary Angioedema
Acronym: BESQAOH
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC21.054
Record Dates: First submitted 2021-04-29; First posted 2021-05-17 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2021-04

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- angiodema hereditary patients: Patient with HAE with or without C1 inhibitor deficiency will respond to an electronic questionnaire
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — electronic questionnaire

SUMMARY:
8 years after the establishment of the therapeutic education program and 14 years after the creation of the National Reference Center for Angioedemas (CREAK), it is necessary to make an inventory in 2021 on the disease experienced by the patient with an assessment the needs and expectations of HAE patients. This assessment would make it possible to see the evolution of these needs and to adjust the price for the overall cost of children and adults in France. It may also allow a comparison of the requests expressed during a similar survey in another French-speaking region such as Quebec.

Main objective is to know the needs and the current satisfaction of the needs, with regard to the disease and the treatment of the targeted patients of hereditary angioedema (HAE)

ELIGIBILITY:
Inclusion Criteria:

* Patient with HAE with or without C1 inhibitor deficiency
* Patient over 15 or parents of a child under 15 with HAE

Exclusion Criteria:

* Patient opposed to the use of their data or refusing to answer the questionnaire
* Adult patients protected by law

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with HAE with or without C1 inhibitor deficiency
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
the needs and the current satisfaction of the needs, with regard to the disease and the treatment of patients with hereditary angioedema (HAE) | baseline
  questionnaire To know the needs and the current satisfaction of the needs, with regard to the disease and the treatment of patients with hereditary angioedema (HAE)

SECONDARY OUTCOMES:
comparaison of results with quebec | baseline
  Comparison of the results of the French questionnaire, only the questions adapted from the Quebec questionnaire, with the results of the Quebec survey conducted by Jean-Nicolas Boursiquot in 2018.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUGA, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided